CLINICAL TRIAL: NCT03893578
Title: First in Human Safety Study of the Synecor Conveyor System Used for Delivery of a Minimally Invasive Mitral Valve
Brief Title: The Conveyor Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Synecor, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYN-FIH-001
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Mitral Valve Insufficiency; Mitral Valve Disease; Mitral Valve Regurgitation; Heart Failure
Keywords: Conveyor System; Sapien 3; cardiovascular disease; TMVR; failing valve; failing bioprosthetic valve
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Failure; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Device: Synecor Conveyor System
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Interventional Arm (Experimental): Access, delivery, and retrieval of the Conveyor system with correct positioning of the valve delivery system to facilitate correct positioning of the implant at the mitral location in patients with a failing bioprosthetic valve.
  Interventions: Device: Mitral valve-in-valve

INTERVENTIONS:
Device: Mitral valve-in-valve — The Synecor Conveyor System shall be used to position the Edwards SAPIEN 3 valve at the mitral location.

SUMMARY:
To demonstrate that the Conveyor System can safely provide left ventricular access to deliver the SAPIEN 3 (Edwards Lifesciences, Irvine, California) transcatheter heart valve in patients who have been diagnosed with prior mitral valve replacement or repair (failing bioprosthetic mitral valve) who are candidates for mitral valve-in-valve procedure.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, multi-center early feasibility study designed to demonstrate that the Conveyor System can safely provide left ventricular access to deliver an Edwards SAPIEN 3 TAVR valve into the mitral valve position in a valve-in-valve procedure. This study will enroll patients with symptomatic heart disease due to a failing bioprosthetic mitral valve (stenosed insufficient, or combined).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able and willing to comply with all assessments in the study.
2. Subject or subjects' legal representative have been informed of the nature of the study, agrees to participate, and has signed the approved consent form.
3. Age of Subject is ≥18.
4. Estimated life expectancy >6 months.
5. Patients demonstrated to have symptomatic post-therapeutic mitral valve dysfunction as determined at diagnostic cardiac catheterization, echocardiography, and/or MR and a mitral valve annulus suitable for a "valve in valve" transcatheter valve replacement procedure using the Edwards SAPIEN 3™ TAVR device based on diagnostic cardiac catheterization, echocardiography and/or MR imaging.
6. Patient has been evaluated by a Heart Team and judged to be a candidate for mitral valve in valve procedure.
7. Patient has femoral and iliac artery dimensions sufficient to accept the study device (>6 mm).
8. Patient is potential surgical candidate.

Exclusion Criteria:

1. Patients with any clinical presentation that will exclude them from receiving a Edwards SAPIEN 3™ percutaneous valve.
2. Patients with vascular disease that would preclude navigation of the Conveyor System.
3. Patients who do not desire to participate in the study.
4. Patients who are judged to be mentally incapable of fully understanding the risks or potential benefits of participation in the study.
5. Patients with visible thrombus in the left atrium or on the mitral valve apparatus/replacement.
6. Patient requires urgent or emergent treatment.
7. Patient has significant aortic valve disease or previous aortic valve replacement.
8. Pregnant patients (must have negative pregnancy test).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Correct Positioning of Implant | 30 Days
  The ability of the Conveyor System to safely position the valve delivery system to facilitate correct positioning of the implant without causing any serious adverse events through 30-day follow up. Cineangiography will be used in delivery to ensure that the implant is orthogonal to the mitral valve annulus and centered within it from multiple views. The patient will be seen in the clinic in a routine follow-up to ascertain any untoward clinical signs or symptoms.